CLINICAL TRIAL: NCT06421948
Title: PI3Kδ Inhibitor Linperlisib Combined With HDAC Inhibitor Chidamide Versus CHOP in Patients With Peripheral T-cell Lymphoma: a Multicenter, Open Label, Phase Ib/II Study
Brief Title: Linperlisib Combined With Chidamide in Patients With PTCL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yanyan Liu (Other Government)
Responsible Party: Sponsor-Investigator, Yanyan Liu, Professor, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYML08
Record Dates: First submitted 2024-05-06; First posted 2024-05-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-05

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cyclophosphamide; Doxorubicin; Epirubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase Ib: Dose-escalation cohort (Experimental): Linperlisib was administered in three dose groups of 40 mg, 60 mg, and 80 mg once daily (QD), with each group enrolling 3-6 patients with newly diagnosed or relapsed/refractory PTCL. Chidamide was given at a fixed dose of 20 mg twice weekly. During the 21-day DLT (dose-limiting toxicity) observation period, the maximum tolerated dose (MTD) of linperlisib was assessed, and the recommended phase II dose (RP2D) was determined for use in the phase II study.
  Interventions: Drug: Linperlisib and chidamide
- Phase IIa: Expansion cohort (Experimental): In newly diagnosed PTCL patients, the efficacy and safety of Linperlisib (RP2D) combined with Chidamide were evaluated. Each treatment cycle is 3 weeks, and patients who responded effectively would receive a total of six cycles of therapy.
  Interventions: Drug: Linperlisib and chidamide
- Phase IIb: Randomized controlled study: experimental arm (Experimental): Patients randomized to the experimental group will receive combination therapy with Linperlisib and Chidamide.
  Interventions: Drug: Linperlisib and chidamide
- Phase IIb: Randomized controlled study: Control arm (Active Comparator): Patients randomized to the control group will receive conventional CHOP or CHOP-like regimen chemotherapy.
  Interventions: Drug: cyclophosphamide, doxorubicin/epirubicin, vincristine, and prednisone

INTERVENTIONS:
Drug: Linperlisib and chidamide — Linperlisib is a selective PI3Kδ inhibitor that has been approved in mainland China for the treatment of relapsed or refractory follicular lymphoma, with a recommended monotherapy dose of 80 mg orally once daily. In this study, Linperlisib was administered at three dose levels of 40 mg, 60 mg, and 80 mg in order to determine the recommended Phase II dose (RP2D) when combined with a fixed dose of Chidamide (20 mg twice weekly).
  Chidamide has been approved in mainland China for the treatment of relapsed or refractory PTCL and double-expressor DLBCL. In this study, it was administered at a fixed dose of 20 mg twice weekly in combination with Linperlisib.
  Arms: Phase Ib: Dose-escalation cohort
Drug: Linperlisib and chidamide — All patients received Linperlisib at the RP2D dose once daily and Chidamide 20 mg twice weekly, with each treatment cycle lasting 3 weeks. After three cycles, an interim efficacy assessment was performed. Patients who showed a therapeutic response received an additional three cycles, and the final efficacy evaluation was conducted after six cycles.
  Arms: Phase IIa: Expansion cohort
Drug: Linperlisib and chidamide — Patients received Linperlisib at the RP2D dose once daily and Chidamide 20 mg twice weekly, with each treatment cycle lasting 3 weeks. After three cycles, an interim efficacy assessment was performed. Patients who showed a therapeutic response received an additional three cycles, and the final efficacy evaluation was conducted after six cycles.
  Arms: Phase IIb: Randomized controlled study: experimental arm
Drug: cyclophosphamide, doxorubicin/epirubicin, vincristine, and prednisone — Patients receive conventional CHOP (or CHOP-like regimens such as CHOPE or EPOCH) chemotherapy, with 3 weeks for one cycle. After three cycles, an interim efficacy assessment was performed. Patients who showed a response received an additional three cycles, and the final efficacy evaluation was conducted after six cycles.
  Arms: Phase IIb: Randomized controlled study: Control arm

SUMMARY:
The phase Ib part of this study aims to determine the recommended phase II dose （RP2D）of linperlisib in combination with chidamide for the treatment of peripheral T-cell lymphoma (PTCL).

The phase IIa part is designed to evaluate the preliminary efficacy and safety of the linperlisib plus chidamide regimen in newly diagnosed PTCL patients.

The phase IIb part compares the efficacy and safety of linperlisib combined with chidamide versus the standard CHOP (CHOP-like) regimen in newly diagnosed PTCL patients.

DETAILED DESCRIPTION:
In the phase Ib trial, participants with newly diagnosed or relapsed/refractory PTCL will receive fixed dose of chidamide (20 mg, twice a week) and escalating dose of linperlisib (40 mg, 60 mg, or 80 mg, once a day), to find out the RP2D.

The phase IIa study is an exploratory efficacy study enrolling newly diagnosed PTCL patients who receive linperlisib in combination with chidamide to evaluate the efficacy and safety of the regimen.

In the phase IIb study, participants with newly diagnosed PTCL will be randomized into experimental arm (arm A) to receive linperlisib in combination with chidamide, or control arm (arm B) to receive standard CHOP (or CHOP-like) regimen chemotherapy.

Interim efficacy assessment will be performed after three cycles of treatment. Responded participants will receive another three cycles of treatment. After a total of 6 cycles of treatment, participants can choose autologous hematopoietic stem cell transplantation, maintenance treatment with linperlisib and/or chidamide, or watch and wait.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years at the time of inclusion (Age 18-80 years for phase Ib and IIa study)
* Patients with a newly diagnosed and histologically confirmed PTCL (phase Ib study includes both newly diagnosed and relapsed/refractory PTCL). Anaplastic large cell lymphoma, NK/T-cell lymphoma, and primary cutaneous T-cell lymphoma are not included.
* ECOG PS 0-2 at protocol entry
* Estimated life expectancy of 6 months or longer
* Measurable disease
* Hemoglobin ≥ 8 g/dL (≥5 mmol/l); Platelets ≥ 75 x 10E9/L; Absolute neutrophil count ≥ 1.0 x 10E9/L; Platelets ≥ 50 x 10E9/L permitted if documented bone marrow involvement; Serum bilirubin ≤ 1.5 x upper limit of normal (ULN); Serum glutamic-oxaloacetic transaminase (AST) and/or serum glutamic-pyruvic transaminase (ALT) ≤ 2.5 x ULN, or ≤ 5 x ULN if elevation is due to hepatic involvement by lymphoma; Serum creatinine ≤ 1.5 x ULNb; left ventricular ejection fraction (LVEF) ≥ 50%
* Women of childbearing potential must use safe anticonception (e.g. contraceptive pills, intrauterine devices etc.) during the study and 12 months after the last administration of study drugs; Male patients must use contraception for the duration of the study and 6 months after the last administration of study drugs if his partner is of childbearing potential
* Written informed consent

Exclusion Criteria:

* Patients previously treated with PI3K inhibitor
* Patients previously treated with chidamide (phase Ib study is not limited by this item)
* Suspected or documented central nervous system involvement by lymphoma
* Patients with positive HIV and/or active hepatitis B and/or hepatitis C infection
* Patients with active, uncontrolled infections
* Unwillingness or inability to comply with the protocol
* Deemed 'unfit' by the treating physician
* Pregnant and/or breastfeeding women
* Concurrent severe and/or uncontrolled medical disease which is not lymphoma-related
* Patients with contraindications to chemotherapy
* Known hypersensitivity to one or more of the study drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Approximately 3 months
  Phase Ib
CRR (Complete response rate) | Through study completion, an average of 3 years
  Phase IIa and IIb

SECONDARY OUTCOMES:
PFS (progression-free survival) | Through study completion, an average of about 3 years
  Phase IIa and IIb
OS | Through study completion, an average of about 3 years
  Phase IIa and IIb
AE (Adverse event) | Through study completion, an average of 3 years
  Phase Ib, IIa and IIb
Physical Functioning and Fatique as Measured by the European Organization for Research and Treatment of Cancer Quality of Life - Core 30 Questionnaire (EORTCQLQ-C30) | Cycle 1 Day 1 through follow-up period
  Phase IIb
Lymphoma Symptoms as Measured by the Functional Assessment of Cancer Therapy -Lymphoma (FACT-Lym) Subscale | Cycle 1 Day 1 through follow-up period
  Phase IIb

OTHER OUTCOMES:
Correlation between baseline tumor gene mutation profile and clinical efficacy (CRR, PFS, OS) | Through study completion, an average of about 3 years
  Phase Ib, IIa and IIb Baseline tumor tissue will be analyzed using a targeted next-generation sequencing (NGS) panel to determine the tumor gene mutation profile, including the presence of predefined somatic mutations. Clinical efficacy will be evaluated by CRR, PFS, and OS as defined in the protocol. The correlations between baseline tumor gene mutation profile and CRR, PFS, and OS will be explored using appropriate statistical methods (Chi-square Test, Fisher's Exact Test, Log-rank, logistic regression, and Cox proportional hazards models).
Correlation between plasma circulating tumor DNA (ctDNA) levels and clinical efficacy (CRR, PFS, OS) | Through study completion, an average of about 3 years
  Plasma circulating tumor DNA (ctDNA) will be measured at baseline and at predefined on-treatment time points using a next-generation sequencing (NGS)-based assay. ctDNA will be quantified as variant allele frequency (VAF, %) and/or copies per milliliter (copies/mL). Clinical efficacy will be evaluated by CRR, PFS, and OS as defined in the protocol. Exploratory analyses will assess the correlations between baseline ctDNA levels, on-treatment ctDNA levels, and changes from baseline in ctDNA, and clinical efficacy outcomes (CRR, PFS, OS) using appropriate statistical methods (Kaplan-Meier Curves, Cox Proportional Hazards Model, Linear Regression Analysis, Generalized Estimating Equations/Mixed Effects Models, Receiver Operating Characteristic [ROC] Curve,Time-dependent Cox Regression Model, Mixed Effects Models, Multiple Comparison Correction, Spearman Rank Correlation, Group Comparisons, and Multivariate Regression Analysis).
Correlation between tumor microenvironment characteristics assessed by single-cell sequencing and clinical efficacy (CRR, PFS, OS) | Through study completion, an average of about 3 years
  Tumor microenvironment characteristics will be assessed using single-cell sequencing or flow cytometry of tumor tissue obtained at baseline (and, if available, at on-treatment time points). Parameters of interest may include the composition and abundance of immune cell subsets (CD8+ T cells, regulatory T cells, NK cell, macrophage subpopulations) and their gene-expression signatures. These variables will be quantified as the proportion of each cell subset among total viable cells (%) or as gene-expression scores. Clinical efficacy will be evaluated by CRR, PFS, and OS as defined in the protocol. The correlations between tumor microenvironment features (e.g., immune cell subset composition and gene-expression-based signatures) and clinical efficacy outcomes (CRR, PFS, OS) will be explored using appropriate statistical methods (Kaplan-Meier Curves, Cox Proportional Hazards Model, Multivariate Cox Regression, Multivariate Logistic Regression, Linear and Logistic Regression......)

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Liu, Principal Investigator — A
Locations (6):
- China (6):
  - Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Liling Zhang, Wuhan, Hubei
  - Yajun Li, Changsha, Hunan
  - Ming Jiang, Chengdu, Sichuan
  - Huilai Zhang, Tianjin, Tianjin Municipality
  - Cong Li, Hangzhou, Zhejiang